CLINICAL TRIAL: NCT05229393
Title: The Effectiveness of Manual Therapy to the Cervical Spine and Diaphragm,Combined With Breathing Reeducation Exercises, in Patients With Non-specific Chronic Neck Pain: A Randomized Controlled Trial
Brief Title: Manual Therapy to the Cervical Spine and Diaphragm Combined With Breathing Reeducation Exercises, in nsCNP Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of West Attica (Other)
Responsible Party: Principal Investigator, Tatsios Petros, Phd cand., MSc, MSc, OMPT, CMP, Clinical Instructor Manual Therapy, University of West Attica
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UWestAttica300921
Record Dates: First submitted 2022-01-27; First posted 2022-02-08 (Actual); Last update posted 2023-11-24 (Actual); Status verified 2023-11

CONDITIONS: Chronic Neck Pain
Keywords: neck pain,diaphragm manual, manual therapy

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Investigator, Outcomes Assessor
Masking Description: the outcome assessor will be blind only for those outcomes that are not self-reported
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Diaphragmatic Manual Therapy Group A (Experimental): Experimental: Diaphragmatic Manual Therapy plus Cervical Manual Therapy plus Breathing Reeducation Exercises group.
  Cervical manual therapy will be the same as for the Manual Control Group (20 minutes).
  Diaphragmatic Manual Therapy (10 minutes) and Breathing Reeducation Exercises (10 minutes). The program will be carried out three times per week lasting four weeks in total. Each session will last about 40 minutes.
  Interventions: Other: Cervical plus Diaphragmatic Manual Therapy plus Breathing Reeducation Exercises
- Cervical Manual Therapy Group B (Sham Comparator): Sham Comparator: Sham Treatment group or Manual Control Group Patients included in this group will receive Cervical Manual Therapy (25 minutes) plus sham Diaphragmatic Manual techniques (15 minutes). The program will be carried out three times per week lasting four weeks in total. Each session will last about 40 minutes.
  Interventions: Other: Cervical Manual Therapy plus sham Diaphragmatic Manual Therapy
- Conventional Physiotherapy Program Group C (Active Comparator): Active Comparator: Conventional Treatment group Patients included in this group will receive a conventional physiotherapy program with Transcutaneous Electrical Nerve Stimulation-TENS (15 minutes) plus Microwave pulsed Diathermy (10 minutes), and soft tissue techniques (15 minutes).
  The program will be carried out three sessions per week during the four weeks. Each session will last about 40 minutes.
  Interventions: Other: Conventional Physiotherapy Program

INTERVENTIONS:
Other: Cervical plus Diaphragmatic Manual Therapy plus Breathing Reeducation Exercises — Diaphragmatic Manual Therapy consists of techniques intended to indirectly stretch and mobilize the diaphragmatic muscle fibers. This will help to improve muscle contraction and decrease tension. The experimental maneuvers include the Doming Diaphragmatic Technique as described by Leon Chaitow, Lewit, and the Manual Diaphragmatic Release Technique as described by Leon Chaitow. Both maneuvers are performed in two sets of 10 repetitions, within a 1-minute interval.
  Cervical Manual Therapy consists of vertebral mobilization techniques according to the Mulligan technique.
  Breathing Reeducation Exercises consist of i) recognition of the abnormal breathing pattern, ii) relaxation techniques for all the primary and accessory respiratory muscles, iii) diaphragm breathing reeducation iv) pursed lips exercise v) reeducation of the normal breathing rate
  Arms: Diaphragmatic Manual Therapy Group A
Other: Cervical Manual Therapy plus sham Diaphragmatic Manual Therapy — Ultrasound sham as Diaphragmatic Manual techniques. Disconnected ultrasound will be applied in the same position as for the experimental group for 15 min as a placebo treatment.
  Cervical Manual Therapy: will consist of vertebral mobilization techniques according to Mulligan -
  Arms: Cervical Manual Therapy Group B
Other: Conventional Physiotherapy Program — Conventional Physiotherapy Program consists of TENS for 15min, Microwave pulsed Diathermy for 10min, soft tissue techniques for 15min
  Arms: Conventional Physiotherapy Program Group C

SUMMARY:
Chronic neck pain (CNP) is reported to be one of the most common musculoskeletal pain syndromes. Studies showed that patients with chronic neck pain compensated with changes in Pain, Function, Musculoskeletal and Respiratory outcomes. The diaphragm is a primary respiratory muscle contributing to postural stability and spinal control. Many studies showed that manual therapy and exercise improve clinical and respiratory outcomes in CNP patients. Few studies highlight the importance of diaphragm manual therapy and Reeducation Breathing Exercises in musculoskeletal diseases and in CNP patients. However, the exact mechanism is still unclear. This study aims to examine the hypothesis that: "Diaphragm Manual Therapy and Breathing Reeducation Exercises combined with cervical manual therapy - improve clinical and respiratory outcomes more than cervical manual therapy intervention only or conventional physiotherapy

DETAILED DESCRIPTION:
Chronic neck pain (CNP) may affect the physical, social, and psychological aspects of the individual, contributing to the increase in costs in society and business. Neck pain is a major cause of morbidity and disability in everyday life and at the workplace, in many different countries and populations, but its basic pathology and pathophysiology are still unclear.

CNP patients present respiratory dysfunction and pain presence is accompanied by a varying amount of decrements in several clinical outcomes affecting the neuromusculoskeletal system like disability, range of motion restriction, and decreased proprioception as well as neuromuscular control. However, the quality of life and psychology of patients with CNP are affected in parallel. The diaphragm is the most important respiratory muscle also contributing to postural stability and spinal control. Several studies have shown that diaphragm manual therapy and breathing retraining exercises can improve respiratory, as well as pain, function, and musculoskeletal outcomes in chronic low back pain. However, the effectiveness in patients with chronic neck pain has not been definitively determined in relation to other physical therapy interventions. The primary purpose of the present study is to determine further the effectiveness of Diaphragmatic Manual Therapy and Breathing Reeducation Exercises in CNP patients. The secondary purpose is to investigate the relationship between CNP, breathing dysfunction, pain, disability, and musculoskeletal clinical outcomes.

The present study is expected to recruit 90 patients with CNP. Patients with CNP will be randomly assigned to (1) Diaphragmatic Manual Therapy plus Cervical Manual Therapy plus Breathing Reeducation Exercises (2) Cervical Manual Therapy plus sham Diaphragmatic Manual Therapy and (3) Conventional Physiotherapy. Each participant will receive a particular intervention program depending on their group allocation. All participants will receive two evaluation sessions before and after the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who have pain for at least 3 months with non-specific mechanical neck pain
* Individuals voluntarily participating in the study
* Patients will also be selected on the basis of demonstrating DB in at least one of a series of tests conducted to assess the extent of their Dysfunctional Breathing (biomechanical, biochemical, psychological)

Exclusion Criteria:

* Pregnancy

  * Contraindications for manual therapy or inability to complete the treatment
  * Patients who received physiotherapy or osteopathic treatment during the last 3 months
  * Individuals with bronchial asthma, chronic bronchitis, emphysema, bronchiectasis and malignancy
  * Medical diagnosis of rheumatologic disease
  * Medical diagnosis of respiratory disease (COPD, asthma)
  * Spine surgery (cervical, spinal, thoracic or abdominal region)
  * Medical diagnosis of cancer (past or present)
  * Whiplash injuries
  * Previous cervical fracture
  * Cervical anatomical changes
  * Thrombotic events, Anaemia or Diabetes
  * Body temperature greater than 37 degrees in the previous 48 hours
  * Obesity (BMI greater than 40)
  * Scoliosis or other diseases that cause spine and chest deformity
  * Positive cervical region instability and positive vertebral artery test
  * Individuals with neurological deficits or with motor loss
  * Individuals who have whiplash injuries, osteoporosis, or rheumatoid disease (such as rheumatoid arthritis, systemic lupus erythematosus, Sjögren's syndrome)

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2022-10-31 (Actual); Primary Completion 2023-11-21 (Actual); Study Completion 2023-11-21 (Actual)

PRIMARY OUTCOMES:
Change in Neck Disability Index (NDI) | change from baseline up to 4 weeks and up to 3 months
  The NDI consists of 10 sections. Each section is scored on a 0 (no pain) to 5 (worst imaginable pain) rating scale. Points summed to a total score. The test can be interpreted as a raw score, with a maximum score of 50, or as a percentage.
Pain Intensity VAS | change from baseline up to 4 weeks and up to 3 months
  Visual Analog Scale: Minimum value = 0 (Best outcome); Maximum value = 100 (Worst Outcome)

SECONDARY OUTCOMES:
Change in Range of motion (ROM) | change from baseline up to 4 weeks and up to 3 months
  A smartphone-based application and KFORCE SENS electronic goniometer, KINVENT, France will be used to accurately measure ROM during neck movements of Flexion-Extension, Left-Right Side Flexion, and Left-Right Rotation.
Craniovertebral Angle | change from baseline up to 4 weeks and up to 3 months
  Lateral Photography- examination of the FHP through lateral photographs can provide very reliable estimates. The reliability remained high in both the sitting and standing position.
Nijmegen Questionnaire (NQ) | change from baseline up to 4 weeks and up to 3 months
  Screening tool used to detect patients with hyperventilation complaints and DB patterns. Scores>20 are used as the cut-score to identify DB in patients with various conditions. NQ values in healthy individuals range from 10 to 12 ± 7 and values do tend to decrease towards these levels after breathing retraining.
Hi-Lo test | change from baseline up to 4 weeks and up to 3 months
  A test that assesses breathing dysfunction. Instructions will be given to the examiners for how to perform and record the Hi-Lo: ''Examiner at the front and slightly to the side of the person have to place one hand on the sternum of the patient and the other hand on their upper abdomen. The examiner has to determine whether thoracic or abdominal motion is dominant during breathing and to what extent this is so. Also, has to check for paradoxical breathing. The extent of thoracic or abdominal breathing rate using a score between 1 and 3.
Single Breath Count (SBC) | change from baseline up to 4 weeks and up to 3 months
  A test that assesses breathing dysfunction. To perform, ask the patient to count out loud after maximal inspiration. The ability to reach 50 indicates normal respiratory function.
End Tidal CO2 (ETCO2) and Respiratory Rate (RR) | change from baseline up to 4 weeks and up to 3 months
  Measured by Capnography. ETCO2 less than 35 mmHg, RR of 16 breaths/min or more, will be considered as signs of respiratory pattern abnormality.
Breath Holding Time | change from baseline up to 4 weeks and up to 3 months
  A test that assesses DB. This test is an indicator of a person's respiratory response to biochemical, biomechanical, and psychological fac-tors, and it seems that abnormally, shortened, BHT may indicate abnormalities in the respiratory function that are closely related to DB. Participants will be instructed to assume a comfortable sitting position and breath usually and gently in and out and at the end of a normal exhalation, they will be asked to pinch their nose and hold their breath. The instruction is to hold their breath until they cannot hold their breath any longer and require breathing in again. According to Kiesel (2020) [30], a BHT <25 secs is con-sidered as a sign of DB.
Chest Expansion | change from baseline up to 4 weeks and up to 3 months
  The difference between the values obtained during deep inspiration and expiration will be determined by tape ruler (cm), high degrees represent better outcome, low degrees represent worse outcome
Hospital and Anxiety Depression Scale (HADS) (Greek version 2007) | change from baseline up to 4 weeks and up to 3 months
  Assesses the level of anxiety and depression experienced by patients in a hospital outpatient clinic. A subscale score >8 denotes anxiety or depression.
Tampa Scale for Kinesiophobia (TSK) (Greek version 2005) | change from baseline up to 4 weeks and up to 3 months
  Kinesiophobia is one of the most frequently employed measures for assessing pain-related fear in pain patients through a 17-item questionnaire.
Adverse events | change from baseline up to 4 weeks and up to 3 months
  Through an interview, potential adverse effects are evaluated during and after the physiotherapy treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Tatsios Petros, Glyfada, Athens, Greece

IPD SHARING:
Plan to Share IPD: Yes
Participant data collected during the trial, after deidentification.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Immediately following publication
Access Criteria: Anyone who wishes to access the data.

REFERENCES:
- [Result] Simoni G, Bozzolan M, Bonnini S, Grassi A, Zucchini A, Mazzanti C, Oliva D, Caterino F, Gallo A, Da Roit M. Effectiveness of standard cervical physiotherapy plus diaphragm manual therapy on pain in patients with chronic neck pain: A randomized controlled trial. J Bodyw Mov Ther. 2021 Apr;26:481-491. doi: 10.1016/j.jbmt.2020.12.032. Epub 2021 Feb 16. PMID 33992285
- [Result] Hwangbo PN, Hwangbo G, Park J, Lee S. The Effect of Thoracic Joint Mobilization and Self-stretching Exercise on Pulmonary Functions of Patients with Chronic Neck Pain. J Phys Ther Sci. 2014 Nov;26(11):1783-6. doi: 10.1589/jpts.26.1783. Epub 2014 Nov 13. PMID 25435700
- [Result] Genebra CVDS, Maciel NM, Bento TPF, Simeao SFAP, Vitta A. Prevalence and factors associated with neck pain: a population-based study. Braz J Phys Ther. 2017 Jul-Aug;21(4):274-280. doi: 10.1016/j.bjpt.2017.05.005. Epub 2017 May 20. PMID 28602744
- [Result] Cieza A, Causey K, Kamenov K, Hanson SW, Chatterji S, Vos T. Global estimates of the need for rehabilitation based on the Global Burden of Disease study 2019: a systematic analysis for the Global Burden of Disease Study 2019. Lancet. 2021 Dec 19;396(10267):2006-2017. doi: 10.1016/S0140-6736(20)32340-0. Epub 2020 Dec 1. PMID 33275908
- [Result] Koseki T, Kakizaki F, Hayashi S, Nishida N, Itoh M. Effect of forward head posture on thoracic shape and respiratory function. J Phys Ther Sci. 2019 Jan;31(1):63-68. doi: 10.1589/jpts.31.63. Epub 2019 Jan 10. PMID 30774207
- [Result] Peng B, Yang L, Li Y, Liu T, Liu Y. Cervical Proprioception Impairment in Neck Pain-Pathophysiology, Clinical Evaluation, and Management: A Narrative Review. Pain Ther. 2021 Jun;10(1):143-164. doi: 10.1007/s40122-020-00230-z. Epub 2021 Jan 12. PMID 33464539
- [Result] Wirth B, Amstalden M, Perk M, Boutellier U, Humphreys BK. Respiratory dysfunction in patients with chronic neck pain - influence of thoracic spine and chest mobility. Man Ther. 2014 Oct;19(5):440-4. doi: 10.1016/j.math.2014.04.011. Epub 2014 Apr 30. PMID 24835338
- [Result] Kapreli E, Vourazanis E, Strimpakos N. Neck pain causes respiratory dysfunction. Med Hypotheses. 2008;70(5):1009-13. doi: 10.1016/j.mehy.2007.07.050. Epub 2007 Oct 23. PMID 17959320
- [Result] Dimitriadis Z, Podogyros G, Polyviou D, Tasopoulos I, Passa K. The Reliability of Lateral Photography for the Assessment of the Forward Head Posture Through Four Different Angle-Based Analysis Methods in Healthy Individuals. Musculoskeletal Care. 2015 Sep;13(3):179-186. doi: 10.1002/msc.1095. Epub 2015 Jan 30. No abstract available. PMID 25640070